CLINICAL TRIAL: NCT01947699
Title: Glycemic Profile in Women With Gestational Diabetes Treated With Glyburide
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI decided to withdrawal study before recruitment started
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Maisa Feghali, Fellow - Maternal Fetal Medicine & Obstetric Pharmacology, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPMC_GLY_GDM
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glyburide once daily (Experimental): Timing of glyburide dosing will be changed, glucose will be monitored using continuous a glucose monitor.
  Interventions: Drug: Glyburide; Device: Continuous glucose monitor
- Glyburide twice daily (Experimental): Dose interval and timing of glyburide dose will be changed, glucose will be monitored using continuous a glucose monitor.
  Interventions: Drug: Glyburide; Device: Continuous glucose monitor
- Mixed meal tolerance test. (Experimental): Subjects will be admitted to the Clinical Translational Research Center, receive a Mixed meal tolerance test and have timed blood draws to assess the effect of glyburide on glucose and insulin metabolism.
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: Glyburide
Device: Continuous glucose monitor
  Arms: Glyburide once daily; Glyburide twice daily

SUMMARY:
Diabetes is more likely to occur during pregnancy. When present only in pregnancy it is called gestational diabetes, and it places both mom and baby at risk for complications. Glyburide is one of the currently used treatments for diabetes during pregnancy. This drug is a medication taken by mouth that decreases sugar levels in the blood. It is known to decrease the risk of complications linked to diabetes in pregnancy. Recent studies in pregnancy have described a difference in the way and how well the drug works compared to when used outside of pregnancy.

Oral blood sugar lowering agents are approved by the Food and Drug Administration (FDA) to lower blood sugar in non-pregnant subjects with diabetes. No oral (taken by mouth) blood-sugar lowering agents are FDA approved for use in pregnancy. Although Glyburide is not FDA approved for this use, it is the most commonly used oral blood sugar lowering agent in pregnancy.

This research study will help us learn more about the variations in blood sugar levels in women with diabetes in pregnancy who are taking glyburide and how changes in the timing of when the glyburide is taken would affect blood glucose levels. The goals of this study are:

* To find the how glucose changes throughout the day in women with diabetes in pregnancy receiving glyburide
* To learn the effect of changing the time of taking glyburide on glucose levels
* To learn the effect of changing the time between glyburide doses on glucose levels
* To see if insulin is secreted the same throughout the day in response to a morning dose of glyburide.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational diabetes
* Singleton gestation
* Receiving glyburide for the treatment gestational diabetes
* Able to give consent

Exclusion Criteria:

* Women who require insulin for the treatment of gestational diabetes
* Diagnosis of pregestational diabetes
* Poor glycemic control, > 50% of blood glucose values over 200mg/dl prior to start of the study
* Women receiving medications that affect glycemic control e.g. steroids, within a week of enrollment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Glucose levels throughout the day | One week

CONTACTS AND LOCATIONS:
Overall Officials: Maisa Feghali, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Hebert MF, Ma X, Naraharisetti SB, Krudys KM, Umans JG, Hankins GD, Caritis SN, Miodovnik M, Mattison DR, Unadkat JD, Kelly EJ, Blough D, Cobelli C, Ahmed MS, Snodgrass WR, Carr DB, Easterling TR, Vicini P; Obstetric-Fetal Pharmacology Research Unit Network. Are we optimizing gestational diabetes treatment with glyburide? The pharmacologic basis for better clinical practice. Clin Pharmacol Ther. 2009 Jun;85(6):607-14. doi: 10.1038/clpt.2009.5. Epub 2009 Mar 18. PMID 19295505
- [Background] Caritis SN, Hebert MF. A pharmacologic approach to the use of glyburide in pregnancy. Obstet Gynecol. 2013 Jun;121(6):1309-1312. doi: 10.1097/AOG.0b013e31829007f0. PMID 23812467